CLINICAL TRIAL: NCT04123886
Title: A Phase I Study Evaluating the Safety, Tolerability and Pharmacokinetics of SCB-313, Recombinant Human Tumor Necrosis Factor-Related Apoptosis-Inducing Ligand-Trimer Fusion Protein, for the Treatment of Malignant Pleural Effusion
Brief Title: A Phase I Study Evaluating SCB-313(Recombinant Human TRAIL-Trimer Fusion Protein) for the Treatment of Malignant Pleural Effusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Clover Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLO-SCB-313-CHN-002
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCB-313 (Experimental)
  Interventions: Drug: SCB-313

INTERVENTIONS:
Drug: SCB-313 — SCB-313 Intrapleural injection, once daily. Single dose on Day 1 in Cycle 0 followed by 7-day safety assessment, then dose on Day 1,2,3 in Cycle 1 followed by 21-day observation .

SUMMARY:
To evaluate the safety and tolerability of single dose of SCB-313 by intrapleural injection.To evaluate the safety and tolerability of repeated dose of SCB-313 by intrapleural injection once a day for 3 days, and to determine the maximum tolerated dose (MTD) of SCB-313.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed cancer of any primary tumor type.
2. Malignant pleural effusion requiring drainage that is histologically or cytologically confirmed;
3. Eastern Cooperative Oncology Group (ECOG) performance status: 0 to 2. Patients with an ECOG performance status of 3 may be included if the Investigator determines that removal of pleural fluid would improve their performance status to 2 or better.
4. Life expectancy of at least 8 weeks.
5. Age ≥18 years and ≤ 75 years;.
6. Body weight ≥45 kg and body mass index ≥17 kg/m2.
7. Adequate hematologic function, defined as:

   1. Platelet count ≥80,000/μL;
   2. Prothrombin time and activated partial thromboplastin time ≤1.5 times the upper limit of normal (ULN);
   3. Absolute neutrophil count ≥1,500 μL;
   4. Hemoglobin ≥8 g/dL (transfusion and erythropoietic agents are allowed). In case there is existence of active bleeding or other persistent condition of either increased destruction or impaired production of erythrocytes, which may require repeated transfusion or erythropoietic treatment, the eligibility must be discussed with the Sponsor on a case by-case basis prior to randomization.
   5. Ablumin≥35g/L
8. Adequate renal function, defined as serum creatinine ≤2.0 times ULN and creatinine clearance >50 mL/minute.
9. Adequate liver function, defined as:

   1. Aspartate aminotransferase and alanine aminotransferase ≤2.0 times ULN for patients without liver metastases, or ≤5 times ULN in the presence of liver metastases;
   2. Bilirubin ≤2.0 times ULN, unless patient has known Gilberts syndrome.
10. Female patients of childbearing potential (excluding women who have undergone surgical sterilization or are menopausal, defined as no menstrual periods for 1 year or more without any other medical reasons) are eligible if they have negative serum pregnancy test result 7 days before the first dose of SCB-313 and are willing to use an effective method of birth control/contraception to prevent pregnancy until 6 months after discontinuation of SCB-313.
11. Both men and women of reproductive potential must agree to use effective contraception during the study and for 6 months after discontinuation of SCB 313.
12. Note: Contraceptive methods that are considered highly effective areas follows: total abstinence, intrauterine device, double barrier method (such as condom plus diaphragm with spermicide), contraceptive implant, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices, or injections with prolonged release), or vasectomized partner with confirmed azoospermia.
13. Willing to attend follow-up visits according to study protocol.

Exclusion Criteria:

1. Significantly loculated pleural effusions not amenable to drainage or patient is unlikely to benefit from intrapleural therapy.
2. Any anti-tumor drug other than the systemic anti-tumor therapy that the subject has stably used and any treatment that may have an effect on the control of pleural effusions. Prior therapy with monoclonal antibody should be stopped per Investigators judgement making sure delayed side effects will not interfere with the DLT evaluation period after SCB-313 therapy.
3. Acute or chronic infection (such as tuberculosis) requiring antiviral or intravenous antibiotics within 2 weeks prior to enrollment.
4. Clinical unstable or uncontrolled concomitant hematologic, cardiovascular, pulmonary, hepatic, renal, pancreatic, or endocrine diseases.
5. History of gross hemoptysis (>2.5 mL) within 3 months prior to enrollment.
6. Residual adverse events (AEs) > Grade 2 from previous treatment.
7. Evidence or suspicion of relevant psychiatric impairment, including alcohol or recreational drug abuse.
8. Myocardial infarction within 6 months prior to treatment and/or prior diagnoses of congestive heart failure (New York Heart Association Class III or IV), unstable angina, unstable cardiac arrhythmia requiring medication, and/or long QT syndrome or QT/QTc interval >450 msec at Baseline.
9. Uncontrolled hypertension defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg confirmed upon repeated measures (note: no more than 3 repeated measures allowed).
10. Major surgery (open procedures) within 4 weeks prior to enrollment.
11. Patient with ileus within 30 days prior to Screening.
12. Positive serology test for human immunodeficiency virus,Syphilis, Hepatitis B virus(HBV) and/or Hepatitis C virus(HCV).
13. Live vaccine within 2 weeks prior to enrollment.
14. Scheduled participation in another clinical study involving an investigational product or device during the DLT observation period of this study.
15. Previous treatment with a TRAIL-based therapy or death receptor 4/5 agonist therapy.
16. Known or suspected hypersensitivity to any component of SCB-313.
17. Any further condition which, in the opinion of the Investigator, may result in undue risk of the patient by participating in the present study.
18. Untreated or uncontrolled central nervous system metastatic disease, leptomeningeal disease, or cord compression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
DLT | 28 days after first dosing
  Dose Limiting Toxicity

SECONDARY OUTCOMES:
AEs | 28 days after first dosing
  Occurrence of adverse events (AEs) and serious adverse events (SAEs)
Immunogenicity | up to 28 days after first dosing
  Occurrence of binding and neutralizing anti-SCB-313 antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospitial, Sichuan University, Chengdu, Sichuan, China